CLINICAL TRIAL: NCT02758990
Title: Interventional Testing of Gene-environment Interactions Via the Verifomics Mobile Application
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting and financial constraints
Sponsor: Verifomics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2016-10

CONDITIONS: Obesity; Rhinitis; Rhinitis, Allergic; Respiratory Sounds; Dyspnea; Headache; Migraine Disorders; Arthritis; Arthralgia; Anxiety; Sleep Initiation and Maintenance Disorders; Sleep Deprivation
Keywords: Food; Nutrigenomics; Precision Medicine; Pharmacogenetics; Lifestyle
MeSH Terms: conditions — Obesity; Rhinitis; Rhinitis, Allergic; Respiratory Sounds; Dyspnea; Headache; Migraine Disorders; Arthritis; Arthralgia; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Sleep Deprivation | interventions — Vitamin A; Tretinoin; Vitamin B 6; Pyridoxine; Ascorbic Acid; Niacinamide; Cholecalciferol; Vitamin E; alpha-Tocopherol; Caffeine; Coffee; Chocolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (24):
- Predictions: BMI vs. Broccoli (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Broccoli
- Predictions: BMI vs. Caffeine (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Caffeine
- Predictions: BMI vs. Coffee (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Coffee
- Predictions: BMI vs. Spinach (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Spinach
- Predictions: BMI vs. Vitamin A (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin A
- Predictions: BMI vs. Vitamin C (Experimental): BMI will be calculated from self-reported weight (once per day) and height (at enrollment). Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin C
- Predictions: Headache vs. Vitamin B6 (Experimental): Headache frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin B6
- Predictions: Headache vs. Vitamin C (Experimental): Headache frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin C
- Predictions: Headache vs. Nicotinamide (Experimental): Headache frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Nicotinamide
- Predictions: Headache vs. Axon Eyewear (Experimental): Headache frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Device: Axon Eyewear
- Predictions: Rhinitis vs Broccoli (Experimental): Rhinitis frequency and severity will be self-reported on a scale from 0 to 10, with 0 indicating no rhinitis, 3 indicating minor rhinitis, 6 indicating rhinitis while preserving the ability to breathe nasally, and 10 indicating rhinitis to such a degree that mouth-breathing is required, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Broccoli
- Predictions: Rhinitis vs Caffeine (Experimental): Rhinitis frequency and severity will be self-reported on a scale from 0 to 10, with 0 indicating no rhinitis, 3 indicating minor rhinitis, 6 indicating rhinitis while preserving the ability to breathe nasally, and 10 indicating rhinitis to such a degree that mouth-breathing is required, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Caffeine
- Predictions: Rhinitis vs Chocolate (Experimental): Rhinitis frequency and severity will be self-reported on a scale from 0 to 10, with 0 indicating no rhinitis, 3 indicating minor rhinitis, 6 indicating rhinitis while preserving the ability to breathe nasally, and 10 indicating rhinitis to such a degree that mouth-breathing is required, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Chocolate
- Predictions: Rhinitis vs Coffee (Experimental): Rhinitis frequency and severity will be self-reported on a scale from 0 to 10, with 0 indicating no rhinitis, 3 indicating minor rhinitis, 6 indicating rhinitis while preserving the ability to breathe nasally, and 10 indicating rhinitis to such a degree that mouth-breathing is required, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Coffee
- Predictions: Rhinitis vs Vitamin A (Experimental): Rhinitis frequency and severity will be self-reported on a scale from 0 to 10, with 0 indicating no rhinitis, 3 indicating minor rhinitis, 6 indicating rhinitis while preserving the ability to breathe nasally, and 10 indicating rhinitis to such a degree that mouth-breathing is required, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin A
- Predictions: Insomnia vs Axon Eyewear (Experimental): Sleep quality will be self-reported about the previous night's sleep on a scale from 0 to 10, with 0 indicating sleep that was not restful at all, 3 indicating mildly restful but insufficient sleep, 6 indicating a functional quality of sleep but not ideal, and 10 indicating ideal sleep, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Device: Axon Eyewear
- Predictions: Insomnia vs Vitamin A (Experimental): Sleep quality will be self-reported about the previous night's sleep on a scale from 0 to 10, with 0 indicating sleep that was not restful at all, 3 indicating mildly restful but insufficient sleep, 6 indicating a functional quality of sleep but not ideal, and 10 indicating ideal sleep, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin A
- Predictions: Insomnia vs Vitamin E (Experimental): Sleep quality will be self-reported about the previous night's sleep on a scale from 0 to 10, with 0 indicating sleep that was not restful at all, 3 indicating mildly restful but insufficient sleep, 6 indicating a functional quality of sleep but not ideal, and 10 indicating ideal sleep, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin E
- Predictions: Insomnia vs Nicotinamide (Experimental): Sleep quality will be self-reported about the previous night's sleep on a scale from 0 to 10, with 0 indicating sleep that was not restful at all, 3 indicating mildly restful but insufficient sleep, 6 indicating a functional quality of sleep but not ideal, and 10 indicating ideal sleep, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Nicotinamide
- Predictions: Insomnia vs Vitamin D3 (Experimental): Sleep quality will be self-reported about the previous night's sleep on a scale from 0 to 10, with 0 indicating sleep that was not restful at all, 3 indicating mildly restful but insufficient sleep, 6 indicating a functional quality of sleep but not ideal, and 10 indicating ideal sleep, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Vitamin D3
- Predictions: Joint pain vs Broccoli (Experimental): Joint pain frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Broccoli
- Predictions: Joint pain vs Caffeine (Experimental): Joint pain frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Dietary Supplement: Caffeine
- Predictions: Joint pain vs Coffee (Experimental): Joint pain frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Coffee
- Predictions: Joint pain vs Spinach (Experimental): Joint pain frequency and severity will be evaluated via a graphical and written pain scale, reported once per day. Each gene-environment interaction of interest will be evaluated to determine its predictive power.
  Interventions: Other: Spinach

INTERVENTIONS:
Dietary Supplement: Vitamin A — Subjects will be asked to increase vitamin A intake by 8000 International Units per day.
  Other Names: Retinol; Retinoic acid
  Arms: Predictions: BMI vs. Vitamin A; Predictions: Insomnia vs Vitamin A; Predictions: Rhinitis vs Vitamin A
Dietary Supplement: Vitamin B6 — Subjects will be asked to increase vitamin B6 intake by 50 mg per day.
  Other Names: Pyridoxine
  Arms: Predictions: Headache vs. Vitamin B6
Dietary Supplement: Vitamin C — Subjects will be asked to increase vitamin C intake by 500 mg per day.
  Other Names: Ascorbic acid
  Arms: Predictions: BMI vs. Vitamin C; Predictions: Headache vs. Vitamin C
Dietary Supplement: Nicotinamide — Subjects will be asked to increase Nicotinamide intake by 500 mg per day.
  Other Names: Niacinamide
  Arms: Predictions: Headache vs. Nicotinamide; Predictions: Insomnia vs Nicotinamide
Dietary Supplement: Vitamin D3 — Subjects will be asked to increase Vitamin D3 intake by 1000 International Units per day.
  Other Names: Cholecalciferol
  Arms: Predictions: Insomnia vs Vitamin D3
Dietary Supplement: Vitamin E — Subjects will be asked to increase vitamin E intake by 400 International Units per day.
  Other Names: α-tocopherol
  Arms: Predictions: Insomnia vs Vitamin E
Other: Broccoli — Subjects will be asked to increase broccoli intake by 8 fluid ounces (~91 grams) per day.
  Other Names: Brassica oleracea
  Arms: Predictions: BMI vs. Broccoli; Predictions: Joint pain vs Broccoli; Predictions: Rhinitis vs Broccoli
Other: Spinach — Subjects will be asked to increase spinach intake by 8 fluid ounces (~30 grams) per day.
  Other Names: Spinacia oleracea
  Arms: Predictions: BMI vs. Spinach; Predictions: Joint pain vs Spinach
Dietary Supplement: Caffeine — Subjects will be asked to increase caffeine intake by taking 200mg caffeine orally once per day.
  Other Names: 1,3,7-Trimethylpurine-2,6-dione
  Arms: Predictions: BMI vs. Caffeine; Predictions: Joint pain vs Caffeine; Predictions: Rhinitis vs Caffeine
Other: Coffee — Subjects will be asked to increase coffee intake by drinking 2 cups (177 mL each) of coffee per day.
  Arms: Predictions: BMI vs. Coffee; Predictions: Joint pain vs Coffee; Predictions: Rhinitis vs Coffee
Device: Axon Eyewear — Subjects will be asked to utilize the therapeutic eyewear when exposed to bright or fluorescent light.
  Arms: Predictions: Headache vs. Axon Eyewear; Predictions: Insomnia vs Axon Eyewear
Other: Chocolate — Subjects will be asked to increase chocolate intake by eating 57g per day.
  Arms: Predictions: Rhinitis vs Chocolate

SUMMARY:
The purpose of this study is to study interactions between genes, lifestyle environmental factors like foods, nutritional supplements and non-invasive medical devices and health factors that can be measured without specialized medical equipment in order to develop lifestyle recommendations tailored to individual genetics for a host of common chronic health conditions.

DETAILED DESCRIPTION:
The study is composed of multiple interventions which will last between 2 and 6 months that evaluate a suite of predictions about the way that a given environmental factor impacts a specific health outcome based on genetic information obtained from direct-to-consumer genotyping providers (AncestryDNA and 23andMe). Substances of interest include foods, nutritional supplements and non-invasive medical devices.

A minimum of 500 subjects will be enrolled in each intervention, and only those subjects which are predicted to benefit from the intervention when considering all sites of interest will be assigned to an intervention. The predictions are based on hundreds to thousands of sites of interest at high minor allele frequency single nucleotide polymorphisms and predictions about response are derived from the aggregate genotype at all loci considered. As such each site of interest will have a built-in negative control group composed of individuals enrolled in the intervention despite a genotype at that site that does not predict a benefit. The rate that each site of interest makes correct predictions about subject response will be compared to randomly-selected sites in order to quantify placebo effects and establish quality metrics for the predictions.

Enrollment and participation are conducted remotely. Participants will upload genetic information from a direct-to-consumer provider through a mobile or web browser application, and informed consent and inclusion/exclusion criteria are accomplished remotely. After the informed consent process, participants are asked what phenotype of interest (weight, migraines, insomnia, etc.) they are interested in studying, their genetic information is evaluated and they are allowed to select an intervention they qualify for based on their genetics that they would like to participate in. Participants then answer a series of questions to establish baseline data on relevant factors as well as evaluate the inclusion and exclusion criteria; participants that qualify for the intervention are then given specific instructions on how to participate, and may then use the software to report data during the intervention. Each intervention utilizes a specific product rather than a general class of product to reduce noise from differing sourcing, distribution, storage and manufacturing practices.

ELIGIBILITY:
Inclusion Criteria:

* For BMI interventions, BMI > 25
* For headache interventions, more than 2 headache-days per month
* For insomnia interventions, at least one day of self-reported poor sleep per week
* For rhinitis interventions, more than 2 days with symptoms per month
* For joint pain interventions, at least one day of self-reported joint pain per week

Exclusion Criteria:

* Women who are pregnant, nursing or attempting to become pregnant
* Immediately life-threatening disease
* Current use of nutritional supplements of interest (excluded from those interventions to prevent overdose)
* For spinach interventions, gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Frequency of correct predictions | Assessed 30 days after enrollment, comparing values of phenotypes of interest in the final week of the intervention to the value at enrollment and determining if the actual response is consistent with the prediction made prior to enrollment
  Each site of interest is being evaluated for its ability to make correct predictions about subject response. This frequency will be compared via a variety of statistical techniques to that expected by chance to establish its clinical utility.

SECONDARY OUTCOMES:
Genotype-independent effects of substances of interest | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
  Baseline responses to environmental factors studied in terms of phenotypes of interest are measured to remove this potential bias from the analysis of predictive power.
Change in body mass index | Assessed 30 days after enrollment, comparing value at enrollment to value after 30 days of participation
Change in headache severity | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in headache frequency | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in rhinitis severity | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in rhinitis frequency | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in insomnia frequency | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in insomnia severity | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in joint pain severity | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
Change in joint pain frequency | Assessed 30 days after enrollment, comparing value at enrollment to value after in the final week of participation
"Question of the day" questionnaire | Daily for the duration of participation (2 to 6 months), starting on the day of enrollment and ending when the intervention is concluded, either because the scientific endpoints are met or the subjects voluntarily halt participation..
  Asynchronous longitudinal observations about subject health, diet, environment, lifestyle and anecdotal observations to be used to guide future studies, control for co-linear changes in behavior, monitor for serendipitous events and assess environment-environment interactions. Subjects are asked to answer one question from the survey per day, and questions are asked recurrently at question-specific intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Brody Holohan, PhD, Principal Investigator — Verifomics LLC
Locations (1):
- Verifomics, LLC, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website that begins the remote enrollment and participation process. Advertising material present on the site has been approved by the institutional review board. — http://verifomics.com/